CLINICAL TRIAL: NCT04717492
Title: An Observational Study of Beta-Blocker Use in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Acute Myocardial Infarction
Brief Title: An Observational Study of Beta-Blocker Use in Patients With COPD and Acute MI
Acronym: BLOCK2
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 1512M81981-Observational
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Cardiac; Cardiovascular; Beta blockers; Acute Myocardial Infarction; Cardiac Catheterization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The study is a prospective, observational study of patients admitted to the BLOCK COPD network hospitals with acute AMI and Chronic Obstructive Pulmonary Disease (COPD) to determine the prevalence of COPD in patients admitted to the hospital with an acute myocardial infarction (AMI) and to characterize the phenotypic expression and severity of their underlying lung disease. Patients with will be identified via the EMR. 571 participants will be enrolled.

DETAILED DESCRIPTION:
Specific Aim 1. To determine the prevalence of COPD in patients admitted to the hospital with an acute myocardial infarction (AMI) and to characterize the phenotypic expression and severity of their underlying lung disease.

Patients admitted to the hospital and who undergo cardiac catheterization for an AMI will be identified through the electronic medical record (EMR). Those with a diagnosis of COPD in the EMR will be offered participation in the study. Baseline characterization will include demographics, smoking history, prior history of exacerbations in the year before admission, supplemental oxygen use, respiratory and cardiac medication use, comorbidities including history of coronary artery disease, heart failure and ejection fraction, and pulmonary function data as available in the EMR. Results of this Aim will provide data about the prevalence and clinical characteristics of COPD in the hospitalized population with AMI in our network. The Aim will also provide an estimate of the number of annual admissions for patients with COPD and AMI.

Specific Aim 2. To determine the association between beta-blocker use at discharge and cardiopulmonary outcomes in patients with COPD and AMI.

Patients with AMI and EMR-documented COPD will be followed, prospectively from the time of discharge using review of the electronic medical record and as local guidance permits, phone calls at 3 and 6 months. The investigators will determine the associations between beta-blocker use at discharge and the risk for all-cause mortality, recurrent ischemic events, and hospitalization for COPD exacerbation adjusting for baseline characteristics and COPD severity.

Because of the coronavirus disease 2019(COVID-19) pandemic and the possibility of limited access to hospitalized patients, the study consists of three options for enrollment. Option 1 or 2 is preferable if local guidance permits.

Option 1: A total of 3 visits including 1 in person visit in the hospital and 2 follow up phone calls with EMR review at 3 and 6 months after discharge. Sites may consider alternatives to in person consent and data collection including by telephone or video conference.

Option 2: EMR review at the time of hospital admission followed by post-discharge telephone consent and 2 follow up phone calls with EMR review at 3 and 6 months.

Option 3: EMR review at the time of hospital admission and follow-up review of the EMR at 3 and 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent (applicable for Option 1 and 2 only)
2. Men and women age 35 or older
3. Admitted to hospital from the Emergency Department or by hospital to hospital transfer with a primary diagnosis of AMI
4. Undergo cardiac catheterization for AMI
5. EMR-documented COPD

Exclusion Criteria:

1. Cognitive disorder that in the judgment of the investigator impairs understanding of the study objectives or assessments (applicable for Option 1 only)
2. Vulnerable populations, including prisoners and pregnant women

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects hospitalized and who undergo cardiac catheterization with AMI and have EMR-documented COPD.
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dransfield, MD, Principal Investigator — University of Alabama at Birmingham; John Connett, PhD, Principal Investigator — University of Minnesota; Stephen Lazarus, MD, Principal Investigator — University of California, San Francisco
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco-Fresno, Fresno, California
  - LA BioMed at Harbor-UCLA Medical Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Louisiana State University, New Orleans, Louisiana
  - University of Maryland Baltimore, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Veteran's Administration Medical Center, Minneapolis, Minnesota
  - HealthPartners Research Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Presbyterian/Queens, Flushing, New York
  - Columbia University, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - The University of Vermont, Burlington, Vermont
  - University of Washington School of Medicine, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to the hospital and who undergo cardiac catheterization for an AMI were identified through the electronic medical record (EMR). Patients with EMR-documented Chronic Obstructive Pulmonary Disease (COPD) that were discharged alive were followed, prospectively from the time of discharge using review of the electronic medical record and as local guidance permitted, phone calls at 3 and 6 months. Comparisons of participants discharged with a beta
Pre-assignment Details: This is an observational study. Participants that were discharged alive were categorized based on whether they had a beta blocker prescription at discharge.
Groups:
- Not Discharged With Beta Blockers: Participants discharged without a beta blocker prescription
- Discharged With Beta Blockers: Participants discharged with a beta blocker prescription
Period: Overall Study
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Started | 77 | 502
Completed | 73 | 480
Not Completed | 4 | 22
Not completed — Withdrawal by Subject | 2 | 13
Not completed — Lost to Follow-up | 2 | 9

BASELINE CHARACTERISTICS:
Population: Patients with COPD who underwent cardiac catheterization for AMI categorized by whether they were discharged with or without a prescription for any beta-blocker.
Groups:
- Total: Total of all reporting groups
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers | Total
Number analyzed (Participants) | 77 | 502 | 579
Age, Continuous [Median (Full Range); unit: years] | 68 [42 to 93] | 70 [38 to 94] | 70 [38 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 208 | 243
  Male | 42 | 294 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 13 | 14
  Not Hispanic or Latino | 75 | 483 | 558
  Unknown or Not Reported | 1 | 6 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 403 | 464
  Black | 11 | 68 | 79
  Other | 1 | 13 | 14
  Unknown | 4 | 18 | 22
BMI [Median (Full Range); unit: kg/m^2] | 27.0 [15.5 to 59.2] | 28.0 [15.1 to 63.0] | 27.7 [15.1 to 63.0]
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 24 | 188 | 212
  Former smoker | 46 | 279 | 325
  Never smoker | 7 | 35 | 42
High blood pressure [Count of Participants; unit: Participants] | 67 | 454 | 521
Hyperlipidemia [Count of Participants; unit: Participants] | 61 | 411 | 472
Coronary artery disease [Count of Participants; unit: Participants] | 41 | 344 | 385
Heart attack [Count of Participants; unit: Participants] | 34 | 243 | 277
Heart failure [Count of Participants; unit: Participants] | 25 | 189 | 214
Percutaneous coronary intervention [Count of Participants; unit: Participants] | 30 | 255 | 285
Coronary artery bypass grafting [Count of Participants; unit: Participants] | 15 | 103 | 118
Peripheral vascular disease [Count of Participants; unit: Participants] | 16 | 120 | 136
Stroke [Count of Participants; unit: Participants] | 17 | 63 | 80
Diabetes mellitus [Count of Participants; unit: Participants] | 32 | 205 | 237
Cirrhosis [Count of Participants; unit: Participants] | 3 | 23 | 26
Asthma [Count of Participants; unit: Participants] | 17 | 87 | 104
Obstructive sleep apnea [Count of Participants; unit: Participants] | 21 | 122 | 143
End stage renal disease [Count of Participants; unit: Participants] | 5 | 33 | 38
Depression [Count of Participants; unit: Participants] | 27 | 123 | 150
Anxiety [Count of Participants; unit: Participants] | 32 | 121 | 153
Cancer [Count of Participants; unit: Participants] | 14 | 110 | 124
Organ transplantation [Count of Participants; unit: Participants] | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of COPD in Patients Admitted to the Hospital With an Acute Myocardial Infarction (AMI)
Description: Results of this Aim will provide data about the prevalence of COPD in the hospitalized population with AMI in our network.
Time Frame: Baseline
Population: Patients who underwent cardiac catheterization for AMI with self-reported or physician-documented COPD and enrolled in the study compared with patients who underwent cardiac catheterization for AMI without self-reported or physician-documented COPD that were screened but not enrolled for follow-up.
  562 participants had COPD out of those screened. Participants were excluded from two sites that screened only patients with COPD.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Who Underwent Cardiac Catheterization for AMI: Patients screened who underwent cardiac catheterization for AMI
Arm/Group | Patients Who Underwent Cardiac Catheterization for AMI
Number analyzed (Participants) | 3458
Participants | 562

2. Primary Outcome: Forced Expiratory Volume (FEV1), L; Post-bronchodilator
Description: Characterize the phenotypic expression and severity of underlying lung disease. Results of this Aim will provide data about the clinical characteristics of COPD in the hospitalized population with AMI in our network.
Time Frame: Baseline
Population: Based on participants with spirometry data available in their medical records in the 3 years prior to their admission.
Measure: Median (Full Range); unit: Liters
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 14 | 83
Liters | 1.6 [0.7 to 2.7] | 1.7 [0.5 to 3.4]

3. Primary Outcome: FEV1 % Predicted; Post-bronchodilator
Description: as for outcome 2
Time Frame: Baseline
Population: Based on participants with spirometry data available in their medical records in the 3 years prior to their admission.
Measure: Median (Full Range); unit: Percent predicted
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 14 | 82
Percent predicted | 51.5 [26.0 to 85.0] | 67.0 [24.0 to 105.0]

4. Primary Outcome: Number of Participants With Prescriptions for Home Oxygen
Description: as for outcome 2
Time Frame: Baseline
Population: Based on participant self report or from electronic medical records if consent not obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 77 | 502
Participants | 16 | 78

5. Primary Outcome: Number of Participants That Received a Course of Systemic Corticosteroids and/or Antibiotics in Past Year
Description: as for outcome 2
Time Frame: Baseline
Population: Based on participant self report or from electronic medical records if consent not obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 77 | 502
Participants | 21 | 111

6. Primary Outcome: Number of Courses of Systemic Corticosteroids and/or Antibiotics in Past Year
Description: as for outcome 2
Time Frame: Baseline
Population: Based on participant self report or from electronic medical records if consent not obtained. Median and range reported based on those who received a course of systemic corticosteroids and/or antibiotics in past year.
Measure: Median (Full Range); unit: COPD exacerbation treatment courses
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 77 | 502
COPD exacerbation treatment courses | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 10.0]

7. Primary Outcome: Respiratory Episodes Requiring Care in the Emergency Department in Past Year
Description: as for outcome 2
Time Frame: Baseline
Population: Based on participant self report or from electronic medical records if consent not obtained.
Measure: Number; unit: episodes
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 77 | 502
episodes | 11 | 69

8. Primary Outcome: Respiratory Episodes Leading to Hospitalization in Past Year
Description: as for outcome 2
Time Frame: Baseline
Population: Based on participant self report or from electronic medical records if consent not obtained.
Measure: Number; unit: episodes
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 77 | 502
episodes | 10 | 56

9. Primary Outcome: Number of Hospitalizations in Past Year
Description: as for outcome 2
Time Frame: Baseline
Population: Based on participant self report or from electronic medical records if consent not obtained. Median and range reported based on those who had respiratory episodes leading to hospitalization.
Measure: Median (Full Range); unit: number of hospitalizations
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 77 | 502
number of hospitalizations | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 15.0]

10. Primary Outcome: Respiratory Episodes Requiring Intubation in Past Year
Description: as for outcome 2
Time Frame: Baseline
Population: Based on participant self report or from electronic medical records if consent not obtained.
Measure: Number; unit: episodes
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 77 | 502
episodes | 0 | 4

11. Primary Outcome: Time to Death, or First Hospitalization or Revascularization Event
Description: Compare the time to death or all-cause hospitalization or revascularization event at 6 months for patients with AMI and COPD who were discharged alive on beta-blockers to that of patients not discharged on beta-blockers.
Time Frame: 6 month follow-up
Population: Based on participant self report if consent obtained and from electronic medical records.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 73 | 480
days | 19 [6 to 64] | 37.5 [14 to 84.25]
Statistical Analysis 1: Comparison: Not Discharged With Beta Blockers vs Discharged With Beta Blockers; Time to death, or first hospitalization or revascularization event was analyzed using cox proportional hazards models with inverse probability of treatment weighting (IPTW) to reduce confounding. Missing data were imputed using multivariate imputation by chained equations with predictive mean matching; Test type: Other; p = 0.962, Regression, Cox — No adjustments for multiplicity were performed; Cox proportional hazard model with inverse probability of treatment weighting as described in primary manuscript; Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.66 to 1.54]

12. Primary Outcome: Risk of Death, Hospitalization or Revascularization Event
Description: Compare the risk of death or all-cause hospitalization at 6 months for patients with AMI and COPD who were discharged alive on beta-blockers to that of patients not discharged on beta-blockers by analyzing number of participants experiencing events. The number of participants will be reported for this outcome.
Time Frame: 6 month follow-up
Population: Based on participant self report if consent obtained and from electronic medical records.
Measure: Count of Participants; unit: Participants
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 73 | 480
Participants | 35 | 195

13. Secondary Outcome: Time to Cardiovascular Disease (CVD) Related Death or First CVD-related Hospitalization/Revascularization Event
Description: Compare the time to first CVD-related event (revascularization, CVD-related hospitalization, or CVD-related death) for patients with AMI and COPD who were discharged alive on beta-blockers to that of patients not discharged on beta-blockers by analyzing number of participants experiencing events and time to first event.
Time Frame: 6 month follow-up
Population: Based on participant self report if consent obtained and from electronic medical records.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 73 | 480
days | 23.5 [9.75 to 97.5] | 37.5 [13 to 97.25]
Statistical Analysis 1: Comparison: Not Discharged With Beta Blockers vs Discharged With Beta Blockers; Time to CVD-related death or hospitalization/revascularization was analyzed using cox proportional hazards models with inverse probability of treatment weighting (IPTW) to reduce confounding. Missing data were imputed using multivariate imputation by chained equations with predictive mean matching; Test type: Other; p = 0.694, Regression, Cox — No adjustments for multiplicity were performed; Cox proportional hazard model with inverse probability of treatment weighting as described in primary manuscript; Cox Proportional Hazard = 1.11, 95% CI 2-sided [0.65 to 1.92]

14. Secondary Outcome: Risk of Cardiovascular Disease (CVD) Related Death or First CVD-related Hospitalization/Revascularization Event
Description: Compare the risk of CVD-related event (revascularization, CVD-related hospitalization, or CVD-related death) for patients with AMI and COPD who were discharged alive on beta-blockers to that of patients not discharged on beta-blockers by analyzing number of participants experiencing events and time to first event.
Time Frame: 6 month follow-up
Population: Based on participant self report if consent obtained and from electronic medical records.
Measure: Count of Participants; unit: Participants
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 73 | 480
Participants | 20 | 114

15. Secondary Outcome: Time to Respiratory/COPD-related Death or Hospitalization Event
Description: Compare the time to respiratory/COPD-related death or hospitalization for patients with AMI and COPD who were discharged alive on beta-blockers to that of patients not discharged on beta-blockers by analyzing the time to first event.
Time Frame: 6 month follow-up
Population: Based on participant self report if consent obtained and from electronic medical records.
Measure: Median (Inter-Quartile Range); unit: dats
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 73 | 480
dats | 93 [17.75 to 114.37] | 61 [37 to 118]
Statistical Analysis 1: Comparison: Not Discharged With Beta Blockers vs Discharged With Beta Blockers; Time to respiratory/COPD-related death or hospitalization was analyzed using Cox proportional hazards models with inverse probability of treatment weighting (IPTW) to reduce confounding. Missing data were imputed using multivariate imputation by chained equations with predictive mean matching; Test type: Other; p = 0.476, Regression, Cox — No adjustments for multiplicity were performed; Cox proportional hazard model with inverse probability of treatment weighting as described in primary manuscript; Cox Proportional Hazard = 0.75, 95% CI 2-sided [0.34 to 1.66]

16. Secondary Outcome: Risk of Respiratory/COPD-related Death or Hospitalization Event
Description: Compare the risk of respiratory/COPD-related death or hospitalization for patients with AMI and COPD who were discharged alive on beta-blockers to that of patients not discharged on beta-blockers by analyzing the number of of participants experiencing events.
Time Frame: 6 month follow-up
Population: Based on participant self report if consent obtained and from electronic medical records.
Measure: Count of Participants; unit: Participants
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
Number analyzed (Participants) | 73 | 480
Participants | 10 | 45

ADVERSE EVENTS:
Time Frame: 6-month followup
Description: Serious Adverse events were classified as any hospitalization after the primary event, or any revascularization. Non-serious adverse events were classified as use of steroids or antibiotics for a respiratory condition or COPD exacerbation.
Arm/Group | Not Discharged With Beta Blockers | Discharged With Beta Blockers
All-Cause Mortality (participants affected / at risk) | 11/73 | 48/480
Serious Adverse Events (participants affected / at risk) | 29/73 | 163/480
Other Adverse Events (participants affected / at risk) | 14/73 | 82/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Not Discharged With Beta Blockers (N=73) | Discharged With Beta Blockers (N=480)
Nonfatal overall hospitalization or revascularization (General disorders) | 29 | 163
Nonfatal CVD hospitalization or revascularization (Cardiac disorders) | 17 | 105
Nonfatal COPD or respiratory hospitalization (Respiratory, thoracic and mediastinal disorders) | 9 | 37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Not Discharged With Beta Blockers (N=73) | Discharged With Beta Blockers (N=480)
Antibiotics or steroids for COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 14 | 82

LIMITATIONS AND CAVEATS:
Relatively small number of patients who were discharged without beta-blockers, which likely limited the power of our study to detect modest differences in outcomes. Only patients who underwent cardiac catheterization were included. Subsequent hospitalization events at facilities outside the BLOCK-COPD network may not have been captured if study staff were not notified of the event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT04717492/Prot_SAP_001.pdf